CLINICAL TRIAL: NCT02173418
Title: The Effect of Phrenic Nerve Blockade on Acute and Chronic Shoulder Pain in Patients for Lobectomy and Pneumonectomy.
Acronym: TOPBLOC
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Region of Southern Denmark (Other); University of Southern Denmark (Other); Læge Fritz Karners og hustrus Foundation (Unknown); Overlæge dr. med. Edgar Schnohr og hustru Gilberte Schnohrs Foundation (Unknown)
Responsible Party: Principal Investigator, Morten Rune Blichfeldt-Eckhardt, Afdelingslæge, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-002844-25; S-20120129 (Other: Regional ethics committee); 2012-002844-25 (EudraCT Number)
Record Dates: First submitted 2014-06-18; First posted 2014-06-25 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Postoperative Pain
Keywords: Postoperative pain; Acute postoperative pain; Chronic postoperative pain; Shoulder pain; Thoracotomy; Thoracoscopy
MeSH Terms: conditions — Pain, Postoperative; Shoulder Pain | interventions — Ropivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ropivacaine (Experimental): Phrenic nerve block with Ropivacaine
  Interventions: Drug: Phrenic nerve block with Ropivacaine
- Placebo (Placebo Comparator): Phrenic nerve block with Sodium chloride
  Interventions: Drug: Phrenic nerve block with saline

INTERVENTIONS:
Drug: Phrenic nerve block with Ropivacaine
  Other Names: Naropin
  Arms: Ropivacaine
Drug: Phrenic nerve block with saline
  Other Names: Sodium Chloride
  Arms: Placebo

SUMMARY:
The purpose of this study was to test whether peroperative infiltration of the phrenic nerve during lung surgery would protect patients against postoperative shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

1. Patients planned for elective lobectomy or pneumonectomy
2. 18 years or more on the day of the operation
3. Danish skills appropriate for fulfilling preoperative questionnaires

Exclusion Criteria:

1. Known contralateral paresis of the Phrenic nerve
2. Allergy to Ropivacaine or Sodium Chloride
3. Preoperative ipsilateral shoulder pain
4. Infection or eczema on the intervention site. Clinical decision
5. Dementia or similar cerebral condition that makes the subject unable to perform a NRS-score of pain. Determined by clinical evaluation
6. Pregnancy
7. Acute porphyria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2012-11; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Shoulder pain within 6 hours after the operation | Retrospective numerical rating scale, 6 hours after the operation
  Shoulder pain 6 hours after the operations. Number of patients and numeric rating scale score (0-10)

SECONDARY OUTCOMES:
Number of patients with shoulder pain during the first 3 postoperative days. | Postoperative days 0-3
NRS for shoulder pain during the first 3 postoperative days. | Postoperative days 0-3
  NRS=numerical rating scale score 0-10
Opioid use during the first 3 postoperative days | Postoperative day 0-3
  Morphine equivalents
Time spent in the recovery room | Measured at discharge from the recovery room. Estimated to be on postoperative day 0 or 1.
Shoulder pain 3 months postoperatively | 3 months postoperatively
NRS for shoulder pain 3 months postoperatively | 3 months postoperatively
  NRS=numerical rating scale 0-10
Thoracic pain 3 months postoperatively | 3 months postoperatively
NRS for thoracic pain 3 months postoperatively | 3 months postoperatively
  NRS=numerical rating scale 0-10
opioid use 3 months postoperatively | 3 months postoperatively
Shoulder function 3 months postoperatively | 3 months postoperatively
  Measured by DASH-score before the operation and after 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Morten R Blichfeldt-Eckhardt, MD, Principal Investigator — Departement of anaesthesia and intensive care, Odense University Hospital, Odense, Denmark
Locations (1):
- Departement of Anaesthesia and intensive care, Odense University Hospital, Odense, Region Syddanmark, Denmark